CLINICAL TRIAL: NCT01815398
Title: Cognitive Skills Training to Improve Vocational Outcome in Homeless Youth
Brief Title: Cognitive Skills Training for Homeless Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #6586; 1R21MH092569-01A1 (NIH)
Record Dates: First submitted 2013-03-13; First posted 2013-03-21 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Affective Disorders; Anxiety Disorders; Attention Deficit Disorder; Substance Abuse
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer skills training (Active Comparator): 26 sessions conducted 2-3 times a week to train in computer skills related to the workforce.
  Interventions: Behavioral: Computer Skills Training
- Cognitive Remediation (Experimental): 26 sessions conducted 2-3 times a week of cognitive remediation
  Interventions: Behavioral: Cognitive Remediation

INTERVENTIONS:
Behavioral: Cognitive Remediation — Neuropsychological Educational Approach to Remediation (NEAR) is an evidence based, manualized cognitive remediation program that targets cognitive deficits (eg memory, processing speed, executive functioning, working memory and attention) with the intent of improving daily functioning.NEAR is conducted in a small group setting, allowing for supportive social interaction while participants work at their own computer station on engaging computerized activities that are selected to address their unique profile of cognitive deficits. Then, as a group they discuss how their respective cognitive activities will help them achieve their vocational goals.
  Other Names: NEAR
  Arms: Cognitive Remediation
Behavioral: Computer Skills Training — Participants utilize an interactive software program that delivers tutorials, lessons, and practice sessions to develop computer skills for office based employment. During the learning activities, the clinician offers coaching and assistance in setting up computerized training exercises as needed.
  Arms: Computer skills training

SUMMARY:
Many young people who are homeless have cognitive deficits which impede their ability to secure and maintain employment. This study looks to see if targeting cognitive deficits can improve cognition and vocational outcome.

DETAILED DESCRIPTION:
The aim of this research is to conduct a controlled study of cognitive remediation, to provide feasibility data on adapting an established empirically-based cognitive intervention for homeless youth to help them attain vocational goals. The ultimate purpose is that youth will improve in cognitive functioning and have better functional outcomes including jobs to sustain independent living.

The results of this study will inform a larger trial on the efficacy of cognitive remediation in homeless youth to improve cognition and vocational outcomes. Hypotheses are that, compared to those in an active control group receiving computerized work-skills training, individuals who receive cognitive remediation will show greater cognitive benefits on proximal measures of neurocognition and evidence better vocational outcome as defined by greater number of hours worked. This study will address the service gap in the use of integrated psychosocial interventions for homeless populations as the first investigation of cognitive remediation in homeless youth.

ELIGIBILITY:
Inclusion Criteria:

* have a current Diagnostic and Statistical Manual (DSM-IV) Axis I diagnosis
* residing at Covenant House New York Rights of Passage Program
* psychiatrically stable for at least 21 days
* English speaking

Exclusion Criteria:

* mental retardation (<70 Intelligence Quotient; IQ) on premorbid intelligence estimate)
* risk for suicide or violence
* unremitted substance dependence within the past 6 weeks

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Global Cognition Score | Baseline, 13, 26 sessions
  A Global Cognition Score will be derived from the average z scores in five domains of cognitive functioning: working memory, verbal memory, processing speed, executive functioning, and attention.

SECONDARY OUTCOMES:
Vocational outcome | Baseline, 13, 26 sessions
  The vocational outcome will be total number of hours worked. Hours worked per week (range of 0 to 40) will be summed from the time of session 1 of cognitive remediation/active control to the time of one month followup.

OTHER OUTCOMES:
Intrinsic Motivation Inventory | Baseline, 13, 26 sessions
  Self-reported motivation for cognitive treatment will be measured using the total score from the Intrinsic Motivation Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Alice A Medalia, PhD, Principal Investigator — Columbia University
Locations (1):
- Covenant House New York, New York, New York, United States

REFERENCES:
- [Derived] Saperstein AM, Lee S, Ronan EJ, Seeman RS, Medalia A. Cognitive deficit and mental health in homeless transition-age youth. Pediatrics. 2014 Jul;134(1):e138-45. doi: 10.1542/peds.2013-4302. PMID 24958581